CLINICAL TRIAL: NCT00840749
Title: International Randomized Study to Compare CyberKnife® Stereotactic Radiotherapy With Surgical Resection in Stage I Non-small Cell Lung Cancer
Brief Title: Randomized Study to Compare CyberKnife to Surgical Resection In Stage I Non-small Cell Lung Cancer
Acronym: STARS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Accuray Incorporated (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARS
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: STARS; Early Stage Non Small Cell Lung Cancer; NSCLC; CyberKnife; Surgery; Accuray
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CyberKnife Stereotactic Radiotherapy (Experimental)
  Interventions: Radiation: CyberKnife Stereotactic Radiotherapy
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Radiotherapy — Central lesion dose/fractionation: 15 Gy x 4 fractions = 60 Gy; Peripheral lesion dose/fractionation: 20 Gy x 3 fractions = 60 Gy
  Other Names: CyberKnife SBRT, CyberKnife SRT, CyberKnife SRS
  Arms: CyberKnife Stereotactic Radiotherapy
Procedure: Surgery — Both open thoracotomy and video assisted thoracotomy (VATS) are acceptable procedures. Surgery may consist of a lobectomy, sleeve resection, bilobectomy or pneumonectomy as determined by the attending surgeon based on the operative findings
  Other Names: Open thoracotomy, video assisted thoracotomy (VATS)
  Arms: Surgery

SUMMARY:
Lung cancer remains the most frequent cause of cancer death in both men and women in the world. Surgical resection using lobectomy with mediastinal lymph node dissection or sampling has been a standard of care for operable early stage NSCLC. Several studies have reported high local control and survival using SBRT in stage I NSCLC patients. SBRT is now an accepted treatment for medically inoperable patients with stage I NSCLC and patients with operable stage I lung cancer are entered on clinical protocols. The purpose of this study is to conduct a phase III randomized study to compare CyberKnife SBRT with surgery, the current standard of care for stage I operable NSCLC.

DETAILED DESCRIPTION:
Objectives:

Primary Goal: To compare overall survival at 3 years.

Secondary goals:

1. To compare disease specific survival at 3 years.
2. To compare 3 year progression free survival at the treated primary tumor site
3. To compare grade 3 and above acute and/or chronic toxicities.
4. To evaluate predictive value of pre and post treatment PET scan in clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of non-small cell cancer will be required by either biopsy or cytology. The following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma with or without BAC features, large cell carcinoma with or without neuroendocrine features, neuroendocrine carcinoma, bronchioloalveolar cell carcinoma, or non-small cell carcinoma not otherwise specified.
2. Eligible patients must have appropriate staging studies identifying them as specific subsets of the revised IASCL state IA or IB based on only one of the following combinations of TNM staging:

   T1, N0, M0 or T2 (<=4 cm), N0, M0
3. A PET/CT scan is required. Patients with hilar or mediastinal lymph nodes with short axis diameter < 1 cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm short axis diameter of hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer. Solitary pulmonary lesions <4 mm will not be considered significant.
4. The patients must be considered a reasonable candidate for surgical resection of the primary tumor. Standard justification for deeming a patient medically operable based on pulmonary function for surgical resection of NSCLC may include any of the following: Baseline FEV1 > 40% predicted, post-operative predicted FEV1 > 30% predicted, diffusion capacity > 40% predicted, absent baseline hypoxemia and/or hypercapnia, exercise oxygen consumption > 50% predicted, absent severe pulmonary hypertension, absent severe cerebral, cardiac, or peripheral vascular disease, and absent severe chronic heart disease.
5. Patients must be ≥ 18 years of age.
6. The patient's Zubrod performance status must be Zubrod 0-2.
7. Mandatory staging studies: Must be done within 8 weeks prior to study entry
8. Patients must sign a study-specific consent form.
9. Patients (men and women) of child bearing potential should use an effective (for them) method of birth control throughout their participation in this study.

Exclusion Criteria:

1. Patients with primary tumors > 4 cm;
2. Patients with well-differentiated neuroendocrine carcinoma (carcinoid tumor)
3. Direct evidence of regional or distant metastases after appropriate staging studies, or synchronous primary or prior malignancy in the past 5 years other than nonmelanomatous skin cancer or in situ cancer;
4. Previous lung or mediastinal radiotherapy;
5. Plans for the patient to receive other concomitant local therapy (including standard fractionated radiotherapy and surgery) while on this protocol except at disease progression;
6. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus;
7. Cannot achieve acceptable SRT planning to meet minimal requirement of target coverage and dose-volume constraints of critical structures (see RT techniques).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Roth, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (19):
- United States (14):
  - Community Regional Medical Center, Fresno, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Denver CyberKnife, Lone Tree, Colorado
  - Jupiter Medical Center, Jupiter, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Parkview Cancer Center, Fort Wayne, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - St. Mary's of Michigan, Saginaw, Michigan
  - St. Mary's Duluth Clinic Health System, Duluth, Minnesota
  - Saint Louis University, St Louis, Missouri
  - St. Mary's, Reno, Nevada
  - St. Luke's Episcopal Hospital, Houston, Texas
  - U.T. M.D. Anderson Cancer Center, Houston, Texas
- China (2):
  - Ruikang Hospital, Nanning, Guangxi
  - Tianjin Cancer Institute and Hospital, Hexi Linchang, Tianjin Municipality
- France (2):
  - Centre Oscar Lambret, Lille
  - Centre Antoine Lacassagne, Nice
- CyberKnife Center of WanFang Medical Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Park S, Kim HJ, Park IK, Kim YT, Kang CH. Stereotactic ablative radiotherapy versus surgery in older patients with stage I lung cancer. Eur J Cardiothorac Surg. 2021 Jul 14;60(1):74-80. doi: 10.1093/ejcts/ezab045. PMID 33668061
- [Derived] Chang JY, Senan S, Paul MA, Mehran RJ, Louie AV, Balter P, Groen HJ, McRae SE, Widder J, Feng L, van den Borne BE, Munsell MF, Hurkmans C, Berry DA, van Werkhoven E, Kresl JJ, Dingemans AM, Dawood O, Haasbeek CJ, Carpenter LS, De Jaeger K, Komaki R, Slotman BJ, Smit EF, Roth JA. Stereotactic ablative radiotherapy versus lobectomy for operable stage I non-small-cell lung cancer: a pooled analysis of two randomised trials. Lancet Oncol. 2015 Jun;16(6):630-7. doi: 10.1016/S1470-2045(15)70168-3. Epub 2015 May 13. PMID 25981812

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CyberKnife Stereotactic Radiotherapy | Surgery
Started | 31 (includes patients who were screened but did not end up treated on protocol) | 27 (includes patients who were screened but did not end up treated on protocol)
Treatment | 20 | 16
1 Month Post tx | 19 | 15
6 Months Post tx | 16 | 10
12 Months Post tx | 14 | 7
18 Months Post tx | 12 | 6
24 Months Post tx | 9 | 3
36 Months Post tx | 1 | 0
Completed | 0 | 0
Not Completed | 31 | 27
Not completed — Death | 1 | 2
Not completed — not treated on study arm | 11 | 11
Not completed — study closed | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CyberKnife Stereotactic Radiotherapy | Surgery | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at evaluation (date of evaluation - date of birth)
  years | 67.5 (10.4) | 67.8 (9.9) | 67.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 7 | 17
ECOG/Zubrod performance status [Number; unit: participants] — patient's level of functioning/quality of daily life
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; cannot carry on any selfcare
  5. - Dead
  participants
    0 | 14 | 12 | 26
    1 | 5 | 4 | 9
    2 | 0 | 0 | 0
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
    Missing | 1 | 0 | 1
Primary Tumour stage [Number; unit: participants] — T stage size/extension of tumor
  T0: No evidence of primary tumor T1a: Melanoma ≤1.0 mm in thickness without ulceration and mitoses < 1/mm 2 T1b: Melanoma ≤1.0 mm in thickness with ulceration or mitoses ≥ 1/mm 2 T2a: Melanomas 1.01-2.0 mm in thickness without ulceration T2b: Melanomas 1.01-2.0 mm in thickness with ulceration
  participants
    T1a | 11 | 10 | 18
    T1b | 5 | 5 | 13
    T2a | 4 | 1 | 5
Lesion Type [Number; unit: participants]
  Peripheral | 16 | 12 | 26
  Central | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The study power was calculated for sample size of 420 patients, enrolled over 7 years. The actual enrollment was 36 patients over 4 years. The study was therefore terminated due to lack of enrollment. The sample size does not allow to analysis of the primary outcome.
  While the study data is not mature enough to evaluate the endpoints of the study, we will attempt to describe the results gleaned from the existing patient population.
Time Frame: 3 years
Population: At the time of study closure, 20 patients were treated on the CyberKnife arm and 16 on the Surgery arm. Two deaths were captured on the Surgery arm during the course of the study and one patient enrolled on the CyberKnife arm passed away before being treated with CyberKnife.
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Stereotactic Radiotherapy | Surgery
Number analyzed (Participants) | 20 | 16
Participants | 19 | 14

2. Post Hoc Outcome: Patient Characteristics
Description: While the study data is not mature enough to evaluate the endpoints of the study, we will attempt to describe the results gleaned from the existing patient population.
Time Frame: 3 years
Population: No patients randomized in either treatment arm made it to 3 years follow-up. No further data was collected or will be collected on the patient population.
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Stereotactic Radiotherapy | Surgery
Number analyzed (Participants) | 20 | 16
Participants
  Pts enrolled at MD Anderson | 12 | 10
  Pts enrolled from other sites | 8 | 6
  Age: 40-49 | 2 | 0
  Age: 50-59 | 1 | 3
  Age: 60-69 | 8 | 8
  Age: 70-79 | 7 | 2
  Age: 80-89 | 2 | 3
  Male | 10 | 7
  Female | 10 | 9
  Central Tumor | 4 | 4
  Peripheral Tumor | 16 | 12
  T1a | 11 | 10
  T1b | 5 | 5
  T2a | 4 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | CyberKnife Stereotactic Radiotherapy | Surgery
All-Cause Mortality (participants affected / at risk) | 1/19 | 2/14
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/16
Other Adverse Events (participants affected / at risk) | 7/20 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyberKnife Stereotactic Radiotherapy (N=20) | Surgery (N=16)
Pulmonary Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — patient experienced Grade 3 pulmonary insufficiency that was coded as "unrelated" to study treatment and secondary to chronic obstructive pulmonary disease (COPD)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — patient was admitted to ICU due to Grade 4 pulmonary embolism, and septic shock secondary to pseudomonas aeruginosa pneumonia, each of these events was coded as "possibly" related to study mandated surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyberKnife Stereotactic Radiotherapy (N=20) | Surgery (N=16)
Chest Wall Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lower Limb Arteritus (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection- sore throat (Infections and infestations) | 1 (1) | 0 (0) — AE reported - sore throat
Rib Fracture (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory Organ System Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No